CLINICAL TRIAL: NCT03862690
Title: A Prospective Non-interventional Study Investigating the Treatment Effect of NovoMix® 30 (Biphasic Insulin Aspart 30) in a Real World Adult Population With Type 2 Diabetes in Algeria
Brief Title: A Research Study, Looking at How NovoMix® Works in People With Type 2 Diabetes in Local Clinical Practice in Algeria
Acronym: B Simple
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-4439; U1111-1208-5168 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Type 2 Diabetes Mellitus: A broad adult population of patients with type 2 diabetes (T2D) requiring insulin therapy in different basal-bolus treatment regimens.
  Interventions: Drug: BIAsp 30

INTERVENTIONS:
Drug: BIAsp 30 — Participants will receive commercially available BIAsp 30 once daily (QD), twice daily (BID) or thrice daily (TID) for 24 weeks according to routine clinical practice. The physician will determine the starting dose and any potential later change to the dose. The decision to switch the patient to NovoMix® 30 is at the treating physician's discretion and independent from the decision to include the patient in the study.
  Other Names: NovoMix®

SUMMARY:
The purpose of the study is to collect information about how NovoMix® 30 works in real world adult population with type 2 diabetes. Participants will get NovoMix® 30 as prescribed by the study doctor. The study will last for about 6-8 months. Participants will be asked questions about their health and their diabetes treatment as part of their study doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* The decision to initiate treatment with commercially available NovoMix® 30 has been made by the patient and the treating physician before and independently from the decision to include the patient in this study
* Male or female, greater than or equal to 19 years at the time of signing informed consent
* Diagnosed with type 2 diabetes and treated with basal insulin plus 1-3 bolus insulin injections per day for at least 24 weeks prior to informed consent
* Available and documented HbA1c value less than or equal to 12 weeks prior to initiation of NovoMix® 30 treatment

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Participation in any clinical trial of an approved or non- approved investigational medicinal product within 24 weeks prior to initiation of NovoMix® 30 treatment. Clinical trials do not include non-interventional studies
* Hypersensitivity to NovoMix® 30 or to any of the excipients
* Pregnancy or intention of becoming pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with type 2 diabetes mellitus, previously treated with basal insulin plus 1-3 bolus insulin injections per day for at least 24 weeks prior to the study,
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-28 (Estimated); Primary Completion 2021-06-28 (Estimated); Study Completion 2021-06-28 (Estimated)

PRIMARY OUTCOMES:
Change in glycosylated haemoglobin A1c (HbA1c) | From baseline (week 0) to end of study (week 24)
  Measured in % point.

SECONDARY OUTCOMES:
Participants achieving HbA1c below 7.0% | At end of study (week 24)
  Number of participants achieving HbA1c less than 7.0% at end of study (week 24) (yes/no).
Particpants achieving HbA1c below 7.5% | At end of study (week 24)
  Number of participants achieving HbA1c less than 7.5% at end of study (week 24) (yes/no).
Partcipants achieving HbA1c below 8.0% | At end of study (week 24)
  Number of participants achieving HbA1c less than 8.0% at end of study (week 24) (yes/no).
Change in rate of severe hypoglycaemia | From baseline (week 0) to end of study visit (as recalled at week 24)
  Measured in episodes/person-year.
Change in total insulin dose | From baseline (week 0) to end of study (week 24)
  Measured in units/day.
Change in Diabetes Treatment Satisfaction (DTSQ) score | From baseline (week 0) to end of study (week 24)
  The DTSQs is a self-completion questionnaire used to assess subject's treatment satisfaction. The DTSQ total score will be based on item 1 and 4-8, which are scored on a scale from 0 to 36, a higher score related to a better perception of treatment satisfaction. Items 2 and 3 will be reported separately on a scale from 0 to 6 as per instruction in the DTSQs manual.
Change in health-related quality of life (EQ-5D) | From baseline (week 0) to end of study (week 24)
  The EQ-5D questionnaire will be used to assess subject's health-related quality of life. This instrument contains 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and measures 5 levels of severity (no problems, slight problems, moderate problems, severe problems and extreme problems). The EQ visual analogue scale (EQ VAS) records the patient's self-rated health on a vertical VAS with scores 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (2):
- Algeria (2):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Constantine

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com